CLINICAL TRIAL: NCT03376945
Title: Safety and Efficacy of n-3 Fatty Acid-based Parenteral Nutrition in Patients With Obstructive Jaundice: A Propensity-matched Study
Brief Title: Application of n-3 Fatty to Patient of Jaundice
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Professor, Huazhong University of Science and Technology
Other Study IDs: Chenxp009
Record Dates: First submitted 2017-12-05; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Obstructive Jaundice; Surgical Procedure, Unspecified
Keywords: n-3; Parenteral nutrition; Jaundice; Propensity score match
MeSH Terms: conditions — Jaundice, Obstructive; Hyperphagia; Jaundice | interventions — TNF-Related Apoptosis-Inducing Ligand

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- trail cohort: n-3 FAs
  Interventions: Drug: trail cohort
- control cohort: Structolipid
  Interventions: Drug: control cohort

INTERVENTIONS:
Drug: trail cohort — Drug: Omega-3 Fatty Acid-Based Parenteral Nutrition Glucose, lipid emulsion, amino acids, fat-and water-soluble vitamins as well as electrolytes were compounded in an "All-In-One" manner. 20% Structolipid and 10% Omegaven (ω-3 fatty acid [FA] mainly; Fresenius-Kabi, Germany) were applied to the trial group, but only Structolipid (ω-6 FA mainly) to the control group for 5 consecutive days postoperatively.
  Other Names: trail
  Groups: trail cohort
Drug: control cohort — Drug: Structolipid Glucose, lipid emulsion, amino acids, fat-and water-soluble vitamins as well as electrolytes were compounded in an "All-In-One" manner. 20% Structolipid and 10% Omegaven (ω-3 FA mainly; Fresenius-Kabi, Germany) were applied to the trial group, but only Structolipid (ω-6 FA mainly) to the control group for 5 consecutive days postoperatively.
  Other Names: control
  Groups: control cohort

SUMMARY:
The safety and efficacy of ω-3 fatty acid in patients with obstructive jaundice is not known. This study provided evidences that ω-3 fatty acid-based parenteral nutrition improved postoperative recovery for patients with obstructive jaundice.

DETAILED DESCRIPTION:
Lipid emulsion enriched in n-3 fatty acid (FA) has been reported to improve postoperative recovery for surgical patients with biliary tract disease, and to improve laboratory and clinical outcomes. The role of it for postoperative patients with jaundice is not clear yet. The object of this research was to evaluate the safety and efficacy of n-3 fatty acid-based parenteral nutrition (PN) for patients with jaundice following Surgical procedure.

This cohort study was a pragmatic, retrospective, single center, matched, clinical trial from May 2014 to June 2017.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of obstructive jaundice must be clear (serum toal bilirubin >51.3umol/L & Imaging evidence), and the obstruction is located in the extrahepatic bile duct;
* Duration of Jaundice is less than 2 weeks;
* Nutritional support is needed
* Nutritional support was administrated during the perioperative period;
* Drainage treatment is effective.

Exclusion Criteria:

* Contraindication for surgical procedure, including Child-Pugh Classification C, severe hemorrhagic disorders, gastrointestinal hemorrhage, acute infectious disease, active phase of chronic hepatitis B & C, severe circulatory disease, renal failure pre -operation, and other unknown cause;
* Abandon treatment;
* Length of stay in hospital <5 day;
* Nutrition support <5 day;
* Conservative treatment;
* Incomplete data;
* Allergic reactions against PN.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort study was a pragmatic, retrospective, single center, matched, clinical trial from May 2014 to June 2017.The trail included obstructive jaundice patients ≥20 years who received PN treatment for ≥5 days for maintenance and improvement of their nutrition status round the operation period. All patients received PN along with the three macronutrients, compounded in an "All-In-One" manner, included amino acids, lipids and glucose, electrolytes, and micronutrients (trace elements and vitamins). The administration was performed with a perfusion pump through a central line within 24 h.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Safety (complications) | postoperative period（1 month ）
  postoperative complications
velocity of the serum total bilirubin clearance | postoperative period（1 month ）
  the velocity of the serum TBIL clearance, which was calculated according to formula behind: (formal TB -TB of current) /time interval

SECONDARY OUTCOMES:
kidney function | postoperative period（1 month ）
  blood test for GFR and creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Doctor, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Hepatic Surgery Center of Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Gong Q, Zhu P, Zhang B, Shu C, Ding Z, Wu J, Zhang B, Chen XP. Safety and efficacy of n-3 fatty acid-based parenteral nutrition in patients with obstructive jaundice: a propensity-matched study. Eur J Clin Nutr. 2018 Aug;72(8):1159-1166. doi: 10.1038/s41430-018-0256-1. Epub 2018 Jul 13. PMID 30006616